CLINICAL TRIAL: NCT04082117
Title: Creating a Culturally-Tailored Intervention to Improve Uptake of Genetic Counseling Among Underserved African American Women With Increased Breast Cancer Risk
Brief Title: Uptake of Genetic Counseling Among African American Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kent F. Hoskins, MD, Associate Professor of Medicine, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-1219
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Risk

STUDY DESIGN:
Intervention Model Description: Educational genetic counseling video
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label (Other): Educational genetic counseling video
  Interventions: Behavioral: Educational video

INTERVENTIONS:
Behavioral: Educational video — Educational genetic counseling video

SUMMARY:
A feasibility study incorporating an educational intervention with cancer genetic risk assessment (CGRA) in the UI Health mammography center

DETAILED DESCRIPTION:
African American (AA) women with a family history of breast cancer who are eligible for genetic counseling and express an interest in participating in the study will be consented and complete a brief survey before and after viewing an educational video on genetic counseling. Survey questions will be read to each participant. The questions capture data on the following constructs regarding genetic counseling: knowledge, attitudes, normative beliefs, motivation, perceived social norms, intention, efficacy beliefs, skills, environmental constraints and opinions on the video. The research team will conduct a review of the UI Health Electronic Medical Record (EMR) 3-6 months after study enrollment to determine if the participant attended a genetic counseling session.

ELIGIBILITY:
Inclusion Criteria:

* African American female age 25-69 years
* Presenting for mammogram at UI Health mammography clinic
* No prior history of breast cancer
* Completed cancer genetic risk assessment (CGRA) in UI Health mammography center
* Recommended for genetic counseling based on CGRA performed at the time of the mammogram.

Exclusion Criteria:

* Unable to complete the informed consent and survey in English
* Previously had genetic counseling for hereditary breast cancer risk
* Prisoners

Ages: 25 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 960 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Knowledge and intentions regarding genetic counseling | 1 hour
  Change in knowledge of genetic counseling and intention to engage in genetic counseling following viewing of educational video based on response to survey designed by study investigators.

SECONDARY OUTCOMES:
Attendance at genetic counseling appointment | 3 months
  Rate that study participants attend a genetic counseling appointment within 3 months of viewing educational video

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hoskins, M.D., Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois Health System, Chicago, Illinois
  - University of Illinois, Chicago, Illinois

REFERENCES:
- [Derived] Henderson V, Madrigal JM, Kendall LC, Parekh P, Newsome J, Chukwudozie IB, Comer-Hagans L, Coffey V, Grumbach G, Spencer S, Rodgers C, Kaur R, Balay L, Maga T, Ramamonjiarivelo Z, Balthazar C, Winn R, Watson K, Odoms-Young A, Hoskins KF. Pilot study of a culturally sensitive intervention to promote genetic counseling for breast cancer risk. BMC Health Serv Res. 2022 Jun 25;22(1):826. doi: 10.1186/s12913-022-08193-x. PMID 35752812